CLINICAL TRIAL: NCT01704729
Title: The Children's WEAR (Wearability and Evaluation of Adjustable Refraction) Trial(Phase 1&2)
Brief Title: The Children's WEAR Trial(Phase 1&2)
Acronym: WEAR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Congdon Nathan, MD,MPH, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: ZOC-WEAR-1
Record Dates: First submitted 2012-09-20; First posted 2012-10-11 (Estimated); Last update posted 2021-03-23 (Actual); Status verified 2021-03

CONDITIONS: Myopia
Keywords: Myopia; Focus groups; refraction; Glasses; spectacles
MeSH Terms: conditions — Myopia | interventions — XRCC4 protein, Arabidopsis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- group2 (Other): Cycloplegic subjective refraction by an experienced optometrist or ophthalmologist
  Interventions: Procedure: group2
- group3 (Other): Cycloplegic subjective refraction by a "vision technician" trained in the Zhongshan Ophthalmic Center's Rural Refractionist Program
  Interventions: Procedure: group3
- group4 (Other): Cycloplegic subjective refraction by an experienced optometrist or ophthalmologist
  Interventions: Procedure: group4
- group1 (Other): Non-cycloplegic self-refraction using First Generation, Child-Specific fluid-filled adjustable spectacles and updated self-refraction protocol
  Interventions: Procedure: group1

INTERVENTIONS:
Procedure: group1 — Non-cycloplegic self-refraction +conventional glasses
  Arms: group1
Procedure: group2 — Cycloplegic subjective refraction by experienced optometrist +conventional glasses
  Arms: group2
Procedure: group3 — Cycloplegic subjective refraction by Rural Refractionist Program + conventional glasses
  Arms: group3
Procedure: group4 — Cycloplegic subjective refraction by an experienced optometrist +ready-made glasses
  Arms: group4

SUMMARY:
Phase I: Focus groups on different designs of adjustable glasses and standard glasses (August-September 2012) Phase II: Two-month randomized trial comparing four groups: (September 2012 - August 2013)

DETAILED DESCRIPTION:
Phase I: Focus groups on different designs of adjustable glasses and standard glasses (August-September 2012) Phase II: Two-month randomized trial comparing four groups: self-refraction with adjustable glasses, receiving custom standard glasses; subjective refraction by an expert refractionist after cycloplegic automated refraction and receiving custom standard glasses; subjective refraction by a rural refractionist after cycloplegic automated refraction, receiving custom standard glasses; and subjective refraction by an expert refractionist after cycloplegic automated refraction receiving ready made glasses (September 2012 - August 2013)

ELIGIBILITY:
Inclusion Criteria:

phase1: - aged 12-17 years

* with <= -1.00D of myopic refractive error in each eye phase2: - 12-15 years old children from two locations in Guangdong Province
* with uncorrected vision </= 6/12 in at least one eye thought to be due to refractive error (that is, correctable to at least 6/7.5 with cycloplegic subjective refraction by an optometrist)

Exclusion Criteria:

* those corrected VA can not up to 6/7.5 with cycloplegic subjective refraction by an optometrist
* those with significant strabismus or vision abnormality (keratopathy, cataract, vitreous macular diseases ), or with vision deficiency ( amblyopia ) children are to be excluded.
* Children developing acquired vision problems other than myopia

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 2300 (Actual)
Dates: Start 2012-09; Primary Completion 2016-04-01 (Actual); Study Completion 2016-04-01 (Actual)

PRIMARY OUTCOMES:
Visual acuity with and without study refractive correction | 2 months

SECONDARY OUTCOMES:
Self-reported and Supplemental visual functioning | 2 months
frequency of glasses-wear and the reason why the frequency is low | 2 months
Accuracy of spectacles given to children | 2 months
Value attached to the glasses and satisfaction to the glasses | 2 months

OTHER OUTCOMES:
Breakage, damage and loss of spectacles | 2 months

CONTACTS AND LOCATIONS:
Overall Officials: Nathan G Congdon, MD,MPH, Principal Investigator — Department of privetive ophthalmology,zhongshan ophthamic center,Sun Yat-sen University
Locations (1):
- Zhongshan Ophthalmic Center, Guangzhou, Guangdong, China